CLINICAL TRIAL: NCT00673361
Title: Phase II Pilot Trial of "Chemo-Switch" Regimen of Biochemotherapy Followed by Daily Low-Dose Temozolomide Plus Sorafenib in Advanced Melanoma
Brief Title: Pilot Trial of "Chemo-Switch" Regimen to Treat Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9361; SR05-888 (Other: Legacy Study ID)
Record Dates: First submitted 2008-05-04; First posted 2008-05-07 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2012-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- "Chemo-Switch" Regimen (Experimental)
  Interventions: Drug: Concurrent decrescendo biochemotherapy regimen; Drug: Low-dose Temozolomide plus Sorafenib

INTERVENTIONS:
Drug: Concurrent decrescendo biochemotherapy regimen — * Temozolomide: 200mg/m^2, daily, PO, days 1-4
  * Vinblastine: 1.5mg/m^2, daily, IV, days 1-4
  * Cisplatin: 20mg/m^2, daily IV, days 1-4
  * IL (interleukin)-2: - 18 milli-International unit (MIU)/m^2, IVCI (intravenous continual infusion), day 1
  * 9 MIU/m^2, IVCI, day 2
  * 4.5 MIU/m^2, IVCI, days 3 & 4
  * Interferon (IFN) alpha: 5 MIU/m^2, daily, SC (subcutaneously), days 1-5
  * 5-day inpatient regimen, to be repeated every 21 days
Drug: Low-dose Temozolomide plus Sorafenib — Temozolomide: 75mg/m^2, PO, QD (quaque die), 6 weeks on/2 weeks off Sorafenib: 400mg, PO, BID, 8 weeks

SUMMARY:
This research study is testing the "chemo-switch" strategy in melanoma, using biochemotherapy initially to shrink tumors and then switching to daily low-dose chemotherapy (temozolomide) together with sorafenib. The purpose of this study is to find out what effects (good and bad) biochemotherapy followed by temozolomide plus sorafenib have on melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed melanoma that is locally advanced or metastatic. Cutaneous, mucosal, ocular, and unknown primary melanoma are all eligible.
* Must have measurable disease, defined by RECIST as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20mm with conventional techniques or >10mm with spiral CT scan.
* May have received prior radiation therapy to one or more non-index lesions (prior radiation to an index lesion is allowable only if progression of the irradiated lesion is demonstrated, with progression defined as an increase of 20% or more in the largest diameter) and/or one prior vaccine therapy for metastatic disease. Prior adjuvant therapy with IFN alpha-2b, vaccine, and/or granulocyte-macrophage colony-stimulating factor (GM-CSF) is permitted. At least 4 weks must have elapsed since the completion of any prior therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients must have normal organ and marrow function as defined below:
* leukocytes >3,000/uL (microliters)
* absolute neutrophil count >1,500/uL
* platelets >100,000/uL
* total bilirubin <2.0mg/dL
* AST (Aspartate transaminase)(SGOT)/ALT (Alanine transaminase)(SGPT) <2.5 X institutional upper limit of normal
* creatinine <1.8mg/dL
* If >50 years of age with one or more cardiac risk factors, must demonstrate normal exercise stress test, stress thallium test, or comparable cardiac ischemia evaluation.
* Must be at least 2 weeks out from major surgery and be free of any active infection requiring antibiotics.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Women must demonstrate a negative pregnancy test prior to initiation of protocol therapy.
* Ability to understand and the willingness to sign a written informed consent form.

Exclusion Criteria:

* Prior chemotherapy, cytokine therapy (including IL-2 or IFN alpha), or antibody therapy for metastatic disease. Prior vaccine therapy is permitted.
* May not be currently receiving any other antineoplastic treatments, including chemotherapy, biologic response modifiers, radiation, vaccine, or investigational agents.
* History of brain metastases.
* Autoimmune disorders that could result in life-threatening complications in the setting of IFN alpha and IL-2 treatment.
* History of sensitivity to E. coli-derived products.
* Concurrent use of corticosteroids or any medical condition likely to require the use of systemic corticosteroids.
* A seizure disorder currently requiring anti-epileptic medication.
* Uncontrolled intercurrent illness including, but not limited to, hypertension, active infection requiring antibiotic therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Evidence of bleeding diathesis.
* Currently on therapeutic anticoagulation. Prophylactic anticoagulation (such as low-dose warfarin) of venous or arterial access devices is allowed provided the PT, PTT (Partial Thromboplastin Time), and international normalized ratio (INR) are normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Morse, M.D., Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | "Chemo-Switch" Regimen
Started | 9
Completed | 7
Not Completed | 2
Not completed — Screen Failure | 2

BASELINE CHARACTERISTICS:
Arm/Group | "Chemo-Switch" Regimen
Number analyzed (Participants) | 9
Age, Customized [Number; unit: participants] — Subjects age 18+
  participants | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Terminated study before accrual goal, no data analysis
Time Frame: 3 weeks, 6 weeks, 16 weeks, & 24 weeks
Arm/Group | Terminated Studybefore Accrual Goal
Number analyzed (Participants) | 0

2. Secondary Outcome: Response Rate as Determined by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Time Frame: post-cycle 1 of low-dose temozolomide plus sorafenib, then every 3 months for up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | "Chemo-Switch" Regimen
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No